CLINICAL TRIAL: NCT01186133
Title: Evaluation of Effectiveness and Safety of the First, Second, and New Drug-Eluting Stents in Routine Clinical Practice
Brief Title: Evaluation of the First, Second, and New Drug-Eluting Stents in Routine Clinical Practice
Acronym: IRIS-DES
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: 2010-035
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Percutaneous Transluminal Coronary Angioplasty
Keywords: coronary disease; drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (27):
- DESSIAN: consecutive patients receiving CYPHER stent
- K-XIENCE: consecutive patients receiving Xience stent
- GENOUS: consecutive patients receiving GENOUS stent
- ELEMENT: consecutive patients receiving PROMUS-ELEMENT stent
- PRIME: consecutive patients receiving XIENCE-PRIME stent
- NOBORI: consecutive patients receiving NOBORI stent
- INTEGRITY: consecutive patients receiving RESOLUTE-INTEGRITY stent
- XPEDITION: consecutive patients receiving XIENCE-XPEDITION stent
- BIOMATRIX: consecutive patients receiving BIOMATRIX stent
- CILOTAX: consecutive patients receiving CILOTAX stent
- DEB: consecutive patients receiving Drug eluting balloon
- DESYNE: consecutive patients receiving DESYNE stent
- PREMIER: consecutive patients receiving PROMUS-PREMIER stent
- ORSIRO: consecutive patients receiving ORSIRO stent
- ONYX: consecutive patients receiving ONYX stent
- BVS: consecutive patients receiving Bioresorbable Vascular Scaffold
- BVS AMI: consecutive acute myocardial infarction patients receiving Bioresorbable Vascular Scaffold
- Ultimaster: consecutive patients receiving Ultimaster stent
- Synergy: consecutive patients receiving Synergy stent
- Biofreedom: consecutive patients receiving Biofreedom stent
- Firehawk: consecutive patients receiving Firehawk stent
- DESyne X2: consecutive patients receiving DESyne X2 stent
- Sierra: consecutive patients receiving Sierra stent
- Tansei: consecutive patients receiving Tansei stent
- Synergy XD and Synergy Megatron™: consecutive patients receiving Synergy XD or Synergy Megatron™ stent
- Xience-Skypoint: consecutive patients receiving Xience-Skypoint stent
- Coroflex ISAR NEO: consecutive patients receiving Coroflex ISAR NEO stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of the new drug-eluting stent (DES), as compared with the first-,second-,third-, and fourth-generation DES, in the "real world" daily practice.

DETAILED DESCRIPTION:
Consecutive patients receiving New DES without a mixture of other DES

ELIGIBILITY:
Inclusion Criteria:

* coronary disease amenable to percutaneous coronary intervention (PCI)
* no clinical and lesion limitations

Exclusion Criteria:

* patients with a mixture of several DES
* terminal illness with life expectancy less than 1 year
* patients with cardiogenic shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients amenable to PCI
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2009-01; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | at 12 months post procedure

SECONDARY OUTCOMES:
Death (all-cause and cardiac) | at 12 months and annually up to 5 years
Myocardial infarction | at 12 months and annually up to 5 years
Stent thrombosis | at 12 months and annually up to 5 years
Target-lesion and target-vessel revascularization | at 12 months and annually up to 5 years
Stroke | at 12 months and annually up to 5 years
Procedural success | at 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, Study Chair — Asan Medical Center
Locations (1):
- Korean centres, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim TO, Kang DY, Ahn JM, Kim MJ, Lee PH, Kim H, Choi Y, Lee J, Lee JM, Jo HH, Park YS, Lim SM, Park SJ, Park DW. Impact of Target Lesion Revascularization on Long-Term Mortality After Percutaneous Coronary Intervention for Left Main Disease. JACC Cardiovasc Interv. 2024 Jan 8;17(1):32-42. doi: 10.1016/j.jcin.2023.10.068. PMID 38199751
- [Derived] Jeong YJ, Hyun J, Lee J, Kim JH, Yang Y, Choe K, Lee JS, Park H, Cho SC, Kang DY, Lee PH, Ahn JM, Park DW, Park SJ; IRIS-DES Registry Investigators. Comparison of Contemporary Drug-Eluting Stents in Patients Undergoing Complex High-Risk Indicated Procedures. JACC Asia. 2022 Mar 1;2(2):182-193. doi: 10.1016/j.jacasi.2021.10.008. eCollection 2022 Apr. PMID 36339122
- [Derived] Yang Y, Hyun J, Lee J, Kim JH, Lee JB, Kang DY, Lee PH, Ahn JM, Park DW, Park SJ; IRIS-DES Registry Investigators. Effectiveness and Safety of Contemporary Drug-Eluting Stents in Patients With Diabetes Mellitus. JACC Asia. 2021 Sep 21;1(2):173-184. doi: 10.1016/j.jacasi.2021.07.009. eCollection 2021 Sep. PMID 36338165
- [Derived] Park S, Ahn JM, Kim TO, Park H, Cho SC, Kang DY, Lee PH, Park DW, Park SJ; IRIS-DES Registry Investigators. Incidence and Impact of Thrombocytopenia in Patients Undergoing Percutaneous Coronary Intervention With Drug-Eluting Stents. Am J Cardiol. 2020 Nov 1;134:55-61. doi: 10.1016/j.amjcard.2020.07.059. Epub 2020 Aug 16. PMID 32891400
- [Derived] Park H, Ahn JM, Kang DY, Lee JB, Park S, Ko E, Cho SC, Lee PH, Park DW, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park SJ. Optimal Stenting Technique for Complex Coronary Lesions: Intracoronary Imaging-Guided Pre-Dilation, Stent Sizing, and Post-Dilation. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1403-1413. doi: 10.1016/j.jcin.2020.03.023. Epub 2020 May 27. PMID 32473888
- [Derived] Lee CH, Ahn JM, Lee KS, Kang DY, Lee PH, Lee SW, Lee CW, Park SW, Park DW, Park SJ; IRIS-DES Registry Investigators. Prevalence, predictors, prognostic significance, and effect of techniques on outcomes of coronary lesion calcification following implantation of drug-eluting stents: a patient-level pooled analysis of stent-specific, multicenter, prospective IRIS-DES registries. Coron Artery Dis. 2021 Jan;32(1):42-50. doi: 10.1097/MCA.0000000000000896. PMID 32310851
- [Derived] Lee CH, Kang DY, Han M, Hur SH, Rha SW, Her SH, Seung KB, Kim KS, Lee PH, Ahn JM, Lee SW, Park SW, Park DW, Park SJ; IRIS-DES Registry Investigators. Differential cutoff points and clinical impact of stent parameters of various drug-eluting stents for predicting major adverse clinical events: An individual patient data pooled analysis of seven stent-specific registries and 17,068 patients. Int J Cardiol. 2019 May 1;282:17-23. doi: 10.1016/j.ijcard.2019.01.108. Epub 2019 Feb 2. PMID 30745256
- [Derived] Lee PH, Kwon O, Ahn JM, Lee CH, Kang DY, Lee JB, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park DW, Park SJ. Safety and Effectiveness of Second-Generation Drug-Eluting Stents in Patients With Left Main Coronary Artery Disease. J Am Coll Cardiol. 2018 Feb 27;71(8):832-841. doi: 10.1016/j.jacc.2017.12.032. PMID 29471933